CLINICAL TRIAL: NCT05955833
Title: 89Zr-DFO*-Trastuzumab PET in Patients With Gastric or Breast Cancer - a Pilot Study
Acronym: HER Image
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82608.018.22
Record Dates: First submitted 2023-06-30; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; HER2-positive Breast Cancer; Gastric Cancer; Metastatic Gastric Cancer; HER2-positive Gastric Cancer
Keywords: PET Imaging; HER2; DFO*; trastuzumab
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-DFO*-trastuzumab PET (Experimental): Patients undergoing the 89Zr-DFO*-trastuzumab PET-scans
  Interventions: Diagnostic Test: 89Zr-DFO*-trastuzumab PET scan

INTERVENTIONS:
Diagnostic Test: 89Zr-DFO*-trastuzumab PET scan — Patients will be administered 37 MBq 89Zr-DFO*-trastuzumab and undergo 3 PET scans on the total body PET scanner at day 1, day 2 and day 4 post-injection (p.i.). The first 3 patients will undergo an additional PET 1-2 h p.i. for dosimetry purposes. Three scans are needed for PK modelling and day 4 p.i. is chosen because it is the same time point as in historical controls. Blood samples for (radioactive) PK analysis will be taken at 10 min, 30 min, 1 h and 2 h p.i., and at every PET scan.

SUMMARY:
The goal of this clinical trial is to test a new PET tracer in patients with HER2-positive breast or gastric cancer. This tracer is made of radioactively labeled trastuzumab, and can show where HER2 is present in the body using a PET-scan. For this research, the investigators make PET-scans in people with HER2-positive, metastasized breast- or gastric cancer. The investigators will investigate if the new HER2-tracer correctly shows all tumor lesions. In the future, this method may be useful to help predict who will benefit from certain HER2-directed therapies.

Participants will be injected with the radioactive tracer once. After injection, participants will undergo 3 PET-scans. Each PET-scan will take a maximum of 60 minutes. The PET-scans are on separate days within a week after injection of the tracer (e.g. 1 day, 2 days and 4 days after injection). Furthermore, the investigators will take 7 blood samples (5 mL each). Participants are not required to stay at the hospital. The first 3 participants will undergo an extra PET-scan 1 - 2 hours after injection.

The amount of radioactivity injected will be 37 MBq (± 10%).

DETAILED DESCRIPTION:
Positron emission tomography (PET) imaging with 89Zr-labeled trastuzumab can potentially discriminate between human epidermal growth factor 2 (HER2) positive and HER2-negative lesions in cancer patients. The obvious advantage over tumor biopsies is that PET imaging provides an overview regarding the heterogeneity of HER2-positivity of all lesions in the patient noninvasively at any given time. The use of a tracer with high specificity and low background signal is critical for accurately identifying positive lesions in patients. Earlier studies in patients with HER2-positive (HER2+) breast cancer and gastric cancer using 89Zr-trastuzumab led to the identification of HER2-positive tumor lesions. However, also lesions were missed and false-positive lesions were seen. Previous work has shown that organs like liver and spleen have significant uptake of 89Zr-trastuzumab. In addition, HER2-directed therapy is most effective in HER2-positive tumors, which are defined as immunohistochemistry (IHC) HER2 expression 3+ or HER2 2+ with gene amplification. Tumors with IHC 0, 1+ or 2+ without amplification are considered HER2-negative. To be able to discriminate between these expression levels with PET imaging, an excellent signal to background ratio is required. Recently, an improved 89Zr-labeled trastuzumab tracer has been developed using a different chelator for 89Zr binding, DFO*, which further improves stability of the 89Zr-labeled trastuzumab tracer. 89Zr-DFO*-trastuzumab preclinically shows improved specificity in uptake of tumor lesions while non-tumor related uptake in bone, liver and spleen is reduced, potentially improving the discrimination of HER2-positive tumor lesions in patients. The investigators hypothesize that the improved 89Zr-DFO*-trastuzumab tracer will lead to a reduced background uptake and thus a better discrimination of HER2-positive tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ breast cancer with metastatic disease starting (new) systemic treatment or
* HER2+ metastatic gastric cancer starting (new) systemic treatment.
* A recent (< 8 weeks of start of study) biopsy confirming HER2+.
* Able to undergo PET imaging procedures.
* At least one lesion of at least 1.5 cm amenable for PET imaging
* Age >18 years of age, willing and able to comply with the protocol as judged by the investigator.
* Signed written informed consent.
* Have a World Health Organisation (WHO) performance status of 0-2.
* Life expectancy of > 3 months.
* Have measurable disease based on RECIST 1.1.
* Adequate organ and bone marrow function, as deemed acceptable by the treating physician
* Women aged <50 years will be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the site.
* Women aged ≥ 50 years will be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago.
* Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP.
* Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP.
* Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.

Exclusion Criteria:

* Contraindications for systemic treatment (as will be assigned by treating physician).
* Pregnant or lactating women.
* Prior allergic reaction to immunoglobulins or immunoglobulin allergy.
* Inability to comply with study procedures.
* Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
89Zr-DFO*-trastuzumab uptake (standard uptake values (SUVmean, %ID/kg) in normal organs/tissues and bloodpool. | SUVmean on day 4 post injection.
89Zr-trastuzumab uptake (standard uptake values (SUVmean, %ID/kg) in normal organs/tissues and bloodpool in historical controls with HER2+ breast cancer (n = 20) who underwent 89Zr-trastuzumab PET imaging. | SUVmean on day 4 post injection.

SECONDARY OUTCOMES:
Tumor uptake: 89Zr-DFO*-trastuzumab uptake (SUV, %ID/kg) in tumor lesions | SUV on day 4 post injection.
Tumor uptake: 89Zr-trastuzumab uptake (SUV, %ID/kg) in tumor lesions in historical controls with HER2+ breast cancer (n = 20) who underwent 89Zr-trastuzumab PET imaging. | SUV on day 4 post injection.
Whole blood pharmacokinetics (PK) of 89Zr-DFO*-trastuzumab (Maximum Plasma Concentration (Cmax) µg/mL) | PK samples are taken at 10, 30, 60 and 120 min post injection, and at 1, 2 and 4 days post injection (at the day of each scan).
Whole blood PK of 89Zr-DFO*-trastuzumab (AUC µg/mL × h) | PK samples are taken at 10, 30, 60 and 120 min post injection, and at 1, 2 and 4 days post injection (at the day of each scan).
Plasma PK of 89Zr-DFO*-trastuzumab (Cmax in µg/mL) | PK samples are taken at 10, 30, 60 and 120 min post injection, and at 1, 2 and 4 days post injection (at the day of each scan).
Plasma PK of 89Zr-DFO*-trastuzumab (AUC µg/mL × h) | PK samples are taken at 10, 30, 60 and 120 min post injection, and at 1, 2 and 4 days post injection (at the day of each scan).
Image-derived PK for 89Zr-DFO*-trastuzumab (µg/mL) | Day 1, 2 and 4 post injection (at each scan)
  For each timepoint, volumes of interest (VOIs) will be delineated in the aorta ascendens, and the activity of the VOI will be calculated afterwards for each timepoint. This calculated activity (in Bq/mL) will then be recalculated to the actual amount of tracer (in µg/mL), which is the image-derived PK.
Literature-derived PK for unlabelled trastuzumab (Cmax in µg/mL) | Day of injection till 7 days post injection.
Literature-derived PK for unlabelled trastuzumab (AUC in µg/mL × day) | Day of injection till 7 days post injection.
Visual PET imaging analysis of tumor uptake of 89Zr-DFO*-trastuzumab and 89Zr-trastuzumab | Day 1, 2 and 4 post injection.
Tumor-to-blood ratio of 89Zr-DFO*-trastuzumab (whole blood and plasma as well as image derived) | Day 1, 2 and 4 post injection.
Tumor-to-image derived blood uptake ratio of 89Zr-trastuzumab | Day 1, 2 and 4 post injection.
HER2 expression measured by IHC on tumor biopsies | The biopsies are at most 8 weeks old at the day of injection, and will be compared with the data of the scans from day 1, 2 and 4 post injection.

CONTACTS AND LOCATIONS:
Overall Officials: C.W. Menke-van der Houven van Oordt, MD, PhD, Principal Investigator — AmsterdamUMC
Locations (1):
- AmsterdamUMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes